CLINICAL TRIAL: NCT03216525
Title: A Randomized, Double-blind, Single-Center Trial of Alvimopan (Entereg) Versus Placebo in Patients Undergoing Radical Cystectomy and Urinary Diversion on an Enhanced Recovery After Surgery ERAS Protocol
Brief Title: Alvimopan Versus Placebo in Patients Undergoing Radical Cystectomy on an Enhanced Recovery Protocol
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mark Preston, Urological Surgeon, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P000330
Record Dates: First submitted 2017-03-13; First posted 2017-07-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — alvimopan

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, single-center double blind trial of Alvimopan versus placebo for improving patient outcomes and cost during radical cystectomy and urinary diversion.
Who Masked: Participant, Investigator
Masking Description: double blind design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Alvimopan (Active Comparator): Oral Alvimopan (Entereg, Merck) 12 mg between 30 minutes and 3 hours before surgery start and twice-daily oral doses postoperatively beginning on day one (AM and PM dosing) until hospital discharge or a maximum of 7 days (15 in-hospital doses).
  Interventions: Drug: Alvimopan
- Matching Placebo (Placebo Comparator): Matching placebo between 30 minutes and 3 hours before surgery start and twice-daily oral doses postoperatively beginning on day one (AM and PM dosing) until hospital discharge or a maximum of 7 days (15 in-hospital doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alvimopan — To determine if Alvimopan during radical cystectomy with urinary diversion results in faster return of bowel function.
  Other Names: Entereg
  Arms: Oral Alvimopan
Drug: Placebo — To determine if placebo during radical cystectomy with urinary diversion results in faster return of bowel function.
  Arms: Matching Placebo

SUMMARY:
To determine if Alvimopan during open or robotic radical cystectomy with urinary diversion results in quicker return of bowel function (GI-2 recovery = time to upper [first toleration of solid food] and lower [first bowel movement] gastrointestinal recovery) compared to placebo.

DETAILED DESCRIPTION:
A prospective, randomized, single-center double blind trial of Alvimopan versus placebo for improving patient outcomes and cost during radical cystectomy and urinary diversion will be performed. A randomized trial is necessary to control for all the known and unknown confounders associated with instituting this novel intervention into a surgical procedure. We will recruit 136 subjects (63 patients in each arm of the study per sample size calculation below, plus additional 10 subjects to account for drop outs). A control group will be administered a placebo in order to directly compare if the Alvimopan intervention is effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radical cystectomy and urinary diversion via open or robotic approach.
* Man or woman between the ages of 18 and 85.
* American Society of Anesthesiologists (ASA) Physical Status Score of class 1-4
* Ileal conduit or ileal neobladder urinary diversion
* Able to understand the study procedures, agreed to participate in the study program, and voluntarily provided informed consent

Exclusion criteria:

* Patients who met any of the following criteria were excluded from participating in the study:
* Scheduled for a partial cystectomy
* Previous total colectomy, gastrectomy, or gastric bypass, or functional colostomy or ileostomy
* More than three doses of opioids (oral or parenteral) within 7 days before the day of surgery
* Chemotherapy for bladder cancer within 1 month of scheduled surgery; prior neoadjuvant chemotherapy allowed.
* Pregnant (identified by a positive serum pregnancy test administered after the initial screening process and before the commencement of study activities) or lactating, or not postmenopausal (no menses for at least 1 year) and of childbearing potential and not using an accepted method of birth control (i.e, surgical sterilization; intrauterine contraceptive device; oral contraceptive, diaphragm, or condom in combination with contraceptive cream, jelly, or foam; or abstinence) (Participants will be asked to use birth control for the entire study and for at least 2 weeks after the last dose of study drug.)
* Participated in another investigational drug or medical device study within 30 days of surgery or planning to be enrolled in another investigational drug or medical device study or any study in which active patient participation was required outside normal hospital data collection during the course of this study
* Clinically significant laboratory abnormalities at screening that would have resulted in the cancellation of surgery
* Using illicit drugs or abusing alcohol
* History of previous surgeries, illness, or behavior (eg, depression, psychosis) that in the opinion of the investigator might have confounded the study results or might have posed additional risk in administering the study procedures
* Patients with severe dementia (as determined from medical records and history. Severe dementia will be defined as dementia that impacts daily functioning.)
* Patients with severe hepatic impairment.
* Patients with end-stage renal disease.
* Patients with heart failure. .
* Patients with complete gastrointestinal obstruction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to Return of Bowel Function | From Day of surgery (Day 0) to Day 30
  To achieve quicker time to return bowel function measured by a composite endpoint of both upper GI recovery (GI-2 recovery = [first toleration of solid food] and lower (first bowel movement) gastrointestinal recovery, taking Alvimopan during radical cystectomy, compared to placebo.

SECONDARY OUTCOMES:
Post-operative Length of Stay | Day of surgery (Day 0) to Day of Discharge (Up to Day 30)
  Post operative LOS was determined by the difference between the date of hospital discharge and the date of surgery; that is the postoperative LOS for a participant was calculated as follows:(date of discharge)-(date of surgery).
Post-operative Morbidity | During hospitalization up to 7 days after surgery
  POM defined as need for nasogastric (NG) tube insertion, hospital stay prolonged because of post-operative ileus (POI) beyond 10 days, or readmission to hospital for POI within 7 days after discharge.
30 Day Complications | Day of surgery (Day 0) to Day 30
  Any Clavien Grade II-V complication.
Readmission to Hospital | Day of Discharge (Up to Day 30)
  Any readmission to hospital for > 24 hours after discharge.
Open vs Robotic Radical Cystectomy | Day of Surgery (Day 0)
  To determine if Alvimopan during open or robotic radical cystectomy with urinary diversion results in decreased time to GI2 recovery
Cost Analysis | Day of surgery (Day 0) to Day 30
  To evaluate costs of surgery and post-operative care between alvimopan and placebo in patients having a radical cystectomy and urinary diversion.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Preston, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Vora AA, Harbin A, Rayson R, Christiansen K, Ghasemian R, Hwang J, Verghese M. Alvimopan provides rapid gastrointestinal recovery without nasogastric tube decompression after radical cystectomy and urinary diversion. Can J Urol. 2012 Jun;19(3):6293-8. PMID 22704317